CLINICAL TRIAL: NCT07124780
Title: Helping Adults With Obsessive-Compulsive Disorder Succeed at Work
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Sapana Patel, Associate Professor of Medical Psychology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NYSPI2025-79; 90IFRE0091 (Other Grant/Funding Number: Administration for Community Living)
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: supported employment; obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Vocational Services plus Cognitive Behavioral Therapy for OCD (Active Comparator): Standard vocational services includes support in finding employment with support from the American Jobs Center over 12 months. Cognitive Behavior Therapy for OCD consists of a standard course of exposure and response prevention over 12 weeks, followed by monthly maintenance sessions for 12 months.
  Interventions: Behavioral: Standard Vocational Services
- Individual Placement and Support plus Cognitive Behavior Therapy for OCD (Experimental): Individual Placement and Support includes support in finding employment with support from an IPS employment specialist over 12 months. Cognitive Behavior Therapy for OCD consists of a standard course of exposure and response prevention over 12 weeks, followed by monthly maintenance sessions for 12 months.
  Interventions: Behavioral: Individual Placement and Support (IPS)

INTERVENTIONS:
Behavioral: Individual Placement and Support (IPS) — Individual Placement and Support is an evidence-based model of supported employment for individuals with mental illness. In IPS, participants will meet with an IPS specialist weekly who will help the study participant create resumes, conduct job searches online or in the community, complete job applications, role-play interviews, and, if requested, accompany them when visiting prospective employers.
  Other Names: IPS
  Arms: Individual Placement and Support plus Cognitive Behavior Therapy for OCD
Behavioral: Standard Vocational Services — In Standard Vocational Services, participants will meet with a representative from the American Jobs Center (AJC) who will help them find a job by identifying their interests, assess their skills and abilities, and advise them on in-demand jobs and potential training opportunities.
  Other Names: SVS
  Arms: Standard Vocational Services plus Cognitive Behavioral Therapy for OCD

SUMMARY:
The purpose of this study is to compare two models of employment services for people with obsessive-compulsive disorder (OCD) interested in finding and maintaining employment. All 40 participants will receive up to 12 sessions of the first-line treatment for OCD called exposure and response prevention, a form of Cognitive Behavioral Therapy (CBT). Assigned by chance, half of the people will also receive Individual Placement and Support (IPS); the other half will receive standard vocational services (SVS). This study will compare these two approaches for helping adults with OCD find and maintain work.

DETAILED DESCRIPTION:
The purpose of this study is to compare two models of employment services for people with obsessive-compulsive disorder (OCD) interested in finding and maintaining employment. In a randomized controlled trial (RCT), we will compare the work and clinical outcomes of individuals with OCD (n=20) who receive CBT plus standard vocational services (SVS) to those who receive this same course of CBT but who also receive Individual Placement and Support (IPS) (n=20). Work and clinical outcomes will be measured before starting CBT, at the end of CBT treatment, and at 6, 9, and 12-month time points.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of OCD
* Currently unemployed and interested in finding competitive employment
* For those currently on medication: On a stable dose of psychiatric medication and willing to remain on this dose for the duration of CBT

Exclusion Criteria:

* Currently receiving supported employment services
* Active suicidality or recent suicide attempt
* Active substance use problem (other than nicotine) that warrants treatment
* Comorbid psychiatric conditions that significantly elevate the risk of study participation
* Reside outside of New York State

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Competitive employment | From enrollment to the end of 12 months
  Employed at least one work shift in an integrated work setting in the open job market at prevailing wages with supervision provided by personnel employed by the business.
Hours worked | From enrollment to the end of 12 months
  Total hours of competitive employment

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (scores range from 0-40 with higher scores indicating greater OCD severity) | From enrollment to the end of 12 months
  Change in severity of OCD symptoms
Quality of Life Enjoyment and Satisfaction Scale (scores range from 14-70 with higher scores indicating greater life satisfaction and enjoyment) | From enrollment to the end of 12 months
  Change in degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning

CONTACTS AND LOCATIONS:
Overall Officials: Sapana R Patel, Ph.D., Principal Investigator — The New York State Psychiatric Institute; Blair Simpson, MD, Ph.D., Principal Investigator — The New York State Psychiatric Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study abstract on National Rehabilitation Information Center — https://www.naric.com/pd-srch-results-rec?search_type=&officer_type=&record_id=4155&load_source=&search_id=469536&start_rec=0&user_name=public.user.929879&load_form=&drill_down=1&filter_id=873